CLINICAL TRIAL: NCT00114218
Title: A Phase II Evaluation of Gemcitabine (NSC #613327) and Docetaxel (NSC # 628503) in the Treatment of Recurrent or Persistent Carcinosarcoma of the Uterus
Brief Title: Gemcitabine and Docetaxel in Treating Patients With Recurrent or Persistent Uterine Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0130E; NCI-2012-02680 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000434843; GOG-0130E (Other: Gynecologic Oncology Group); GOG-0130E (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2014-12

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — Gemcitabine; Docetaxel

ARMS (1):
- Treatment (gemcitabine hydrochloride, docetaxel) (Experimental): Patients receive gemcitabine IV over 30 minutes followed by docetaxel IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Docetaxel

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdC; dFdCyd
Drug: Docetaxel — Given IV
  Other Names: TXT

SUMMARY:
This phase II trial is studying how well giving gemcitabine together with docetaxel works in treating patients with recurrent or persistent uterine cancer. Drugs used in chemotherapy, such as gemcitabine and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the antitumor activity of gemcitabine and docetaxel in patients with recurrent or persistent uterine carcinosarcoma.

II. Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: This is a non-randomized, multicenter study. Patients receive gemcitabine IV over 30 minutes followed by docetaxel IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study within 1-4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed uterine carcinosarcoma

  * Malignant mixed Müllerian tumor, homologous or heterologous type
  * Recurrent or persistent disease

    * Progressive disease after prior local therapy
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * At least 1 target lesion
  * Tumors within a previously irradiated field are not considered target lesions except documented progression or biopsy to confirm persistence at least 90 days after completion of radiation therapy
* Received 1, and only 1, prior chemotherapy regimen for carcinosarcoma

  * Initial treatment may have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
* Ineligible for higher priority GOG protocol (i.e., any active phase III GOG protocol for the same patient population)
* Performance status - GOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No severe pulmonary disease requiring oxygen supplementation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No neuropathy (sensory or motor) > grade 1
* At least 3 weeks since prior biologic therapy or immunotherapy for the malignancy
* No more than 1 prior non-cytotoxic (biologic or cytostatic) regimen (e.g., monoclonal antibodies, cytokines, or small molecule inhibitors of signal transduction) for recurrent or persistent disease
* Recovered from prior chemotherapy
* No more than 1 prior cytotoxic chemotherapy regimen, either as a single agent or combination therapy
* No prior docetaxel or gemcitabine
* At least 1 week since prior hormonal therapy for the malignancy
* Concurrent hormone replacement therapy allowed
* Recovered from prior radiotherapy
* Recovered from prior surgery
* At least 3 weeks since other prior therapy for the malignancy
* No prior cancer treatment that would preclude study therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-03; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Miller, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on March 7, 2005 and was closed to accrual on October 29, 2007
Period: Overall Study
Arm/Group | Treatment (Gemcitabine Hydrochloride, Docetaxel)
Started | 28
Completed | 24
Not Completed | 4
Not completed — Wrong Cell Type | 2
Not completed — Wrong Primary | 1
Not completed — Never Treated | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Gemcitabine Hydrochloride, Docetaxel)
Number analyzed (Participants) | 24
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 2
  50-59 years | 5
  60-69 years | 12
  70-79 years | 4
  >79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Objective Tumor Response Rate (Either Complete Response (CR) or Partial Response (PR) Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesions for measurable disease every other cycle for the first 6 months; every 6 months thereafter until disease progression for up to 5 years.
Population: Eligible and Treated patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (Gemcitabine Hydrochloride, Docetaxel)
Number analyzed (Participants) | 24
Percentage of participants | 8 [1 to 27]

2. Primary Outcome: Incidence of Adverse Effects That Are Grade 3 or Greater as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Description: Count of participants with Toxicities maximum grade greater than or equal to grade 3
Time Frame: Assessed every 28 days (28 days=1 cycle) while on study treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Population: Eligible and Treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Gemcitabine Hydrochloride, Docetaxel)
Number analyzed (Participants) | 24
Participants | 18

ADVERSE EVENTS:
Time Frame: AEs were assessed every 28 days (1cycle) while on study treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | Treatment (Gemcitabine Hydrochloride, Docetaxel)
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Gemcitabine Hydrochloride, Docetaxel) (N=24)
Pain: Extremity-Limb (General disorders) | 1
Pain -Back (General disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Bilirubin (Investigations) | 1
Alkaline Phosphatase (Investigations) | 1
Death No CTCAE Term-Sudden Death (General disorders) | 2
Fatigue (General disorders) | 2
Death No CTCAE Term -Disease Progression NOS (General disorders) | 2
Hemorrhage, GI - Liver (Hepatobiliary disorders) | 1
Abdominal Pain NOS (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema: Limb (General disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 1
Muscle Weakness - Whole body/Generalized (General disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction, GI-Small Bowel (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1
Pain: Kidney (General disorders) | 1
Obstrusction, GU -Ureter (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Gemcitabine Hydrochloride, Docetaxel) (N=24)
Leukopenia (Blood and lymphatic system disorders) | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 18
Anemia (Blood and lymphatic system disorders) | 20
Nausea (Gastrointestinal disorders) | 11
Other Gastrointestinal (Gastrointestinal disorders) | 14
Genitourinary (Renal and urinary disorders) | 2
Neurotoxicity (Nervous system disorders) | 6
Pain (General disorders) | 4
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3
Cardiovascular (Cardiac disorders) | 2
Fatigue (General disorders) | 9
Metabolic (Metabolism and nutrition disorders) | 9
Dermatologic (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 10
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1
SGOT (Investigations) | 3
Alkaline Phosphatase (Investigations) | 3
Lymphatics (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less